CLINICAL TRIAL: NCT03388983
Title: The Effectiveness of Prehabilitation for Patients Undergoing Lumbar Spinal Stenosis: A Randomized Clinical Trial
Brief Title: Effectiveness of Prehabilitation for Patients Undergoing Lumbar Spinal Stenosis Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Université du Québec à Trois-Rivières (Other); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Arnold Wong Yu Lok, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20171204001
Record Dates: First submitted 2017-12-23; First posted 2018-01-03 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Lumbar Spinal Stenosis; Prehabilitation
Keywords: Prehabilitation; Physical activity; Lumbar decompression surgery; Randomized controlled trial
MeSH Terms: conditions — Spinal Stenosis; Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: A single-blinded randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The orthopedic surgeons, outcome assessor and statistician will be blinded to the group allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-week prehabilitation group (Experimental): 6-week prehabilitation
  Interventions: Other: 6-week prehabilitation
- Control group (No Intervention): Patients will receive standard preoperative care (including information about the surgery from an orthopedic surgeon, and a pamphlet summarizing tips of maintaining proper posture and staying active). The usual postoperative care does not include routine rehabilitation program though a short course of rehabilitation may be given based on orthopedic surgeons' discretion.

INTERVENTIONS:
Other: 6-week prehabilitation — Participants will be trained at 3 sessions/week for 6 weeks before the surgery to enhance the overall muscle strength, endurance and spinal stability. A physiotherapist/physical trainer in the participating hospital will supervise the preoperative training. The 45-minute exercise regime will include warm-up and cool-down exercises, and a cardiovascular training on a stationary bicycle, stabilization exercises with emphasis on co-contraction of abdominal and back muscles, and hip raise and hip abduction exercises. The number of repetitions and sets of each exercise will be determined based on individual's ability. Each exercise will be slightly modified based on individual progress. The exercise intensity and complexity will be increased over time.
  Arms: 6-week prehabilitation group

SUMMARY:
Lumbar spinal stenosis (LSS) is a common spinal disease that leads to pain and disability. LSS is defined as lower extremity and perineal symptoms (e.g. intermittent neurogenic claudication/numbness) that may occur with or without low back pain and that is attributed to congenital or acquired narrowing of space available for the neural and vascular tissues in the lumbar spine. Patients with LSS,who do not respond to conservative treatments after 3 months or more, will be eligible for spinal decompression surgery in order to improve functional outcomes.

While various studies have shown that preoperative exercises (prehabilitation) may benefit patients receiving different surgeries (e.g, abdominal surgery, anterior cruciate ligament reconstruction), little is known regarding the effect of prehabilitation for patients undergoing LSS surgery.

The aim of the current randomized controlled trial is to compare the effectiveness of a 6-week prehabilitation program with usual preoperative care in improving multiple outcomes of patients undergoing LSS surgery at baseline, 6 weeks after baseline evaluation, and at 3 and 6 months postoperatively. It is hypothesized that prehabilitation will yield significantly better pre- and post-operative clinical outcomes as compared to usual preoperative care.

DETAILED DESCRIPTION:
Lumbar spinal stenosis (LSS) is a common spinal disease that leads to pain and disability. LSS is defined as lower extremity and perineal symptoms (e.g. intermittent neurogenic claudication/numbness) that may occur with or without low back pain and that is attributed to congenital or acquired narrowing of space available for the neural and vascular tissues in the lumbar spine. Clinical symptoms of LSS include pain, numbness, weakness and warmth in bilateral/unilateral buttock or legs that is precipitated by walking or prolonged standing but is alleviated by sitting or forward bending.

Acquired (degenerative) LSS is the most common degenerative conditions that leads to spinal surgery in adults aged 65 years or older.[2] It is known that the occurrence of degenerative LSS increases with age. Given the aging of the global population (including Hong Kong), the prevalence of degenerative LSS is expected to increase. Major causes of degenerative LSS in older adults are the compression and/or ischemia of nerve roots in diminished lateral or central spinal canals secondary to lumbar spondylosis, progressive hypertrophy of ligamentous/osteocartilaginous structures, or degenerative spondylolisthesis. When patients fail to improve after conservative treatments, surgical intervention is recommended for symptomatic LSS. While decompressive laminectomy/laminotomy with or without spinal fusion for LSS has shown significantly less leg symptoms than conservative treatments, up to 40% of patients undergoing LSS surgery were unsatisfied with the postoperative neurogenic claudication and/or radicular leg symptoms. Accordingly, evidence-based management is needed for patients undergoing LSS surgery to optimize patients' recovery.

Various studies have shown that preoperative exercises (prehabilitation) may benefit patients receiving different surgeries (e.g, abdominal surgery, anterior cruciate ligament reconstruction). Although there is a paucity of prehabilitation for patients undergoing LSS surgery. the potential benefits of prehabilitation substantiate the investigation of prehabilitation for patients undergoing LSS surgery.

Given the above, the aim of the current randomized controlled trial is to compare the effectiveness of a 6-week prehabilitation program with usual preoperative care in improving multiple outcomes of patients undergoing LSS surgery at baseline, 6 weeks after baseline evaluation, and at 3 and 6 months postoperatively. It is hypothesized that prehabilitation will yield significantly better pre- and post-operative clinical outcomes as compared to usual preoperative care.

ELIGIBILITY:
Inclusion Criteria:

* signs of neurogenic claudication
* radiological signs of degenerative LSS on magnetic resonance images or computed tomography images
* radiculopathy with or without low back pain for more than 3 months that is unresponsive to conservative intervention
* Oswestry Disability Index (ODI) > 30 out of 100
* patients undergoing open or minimally invasive laminotomy/laminectomy
* willing to complete pre- and post-operative questionnaires and physical assessments at prescheduled time points

Exclusion Criteria:

* inability to read, speak and understand English/Chinese
* inability to give informed consent
* surgical management for lumbar fractures, tumors, synovial cysts, and scoliosis correction
* any revision lumbar spine surgery, (5) diagnosis of chronic pain conditions (e.g. fibromyalgia)
* presence of a neurological or systematic neuromuscular diseases (e.g. multiple sclerosis, stroke, or rheumatoid arthritis)
* planning for spinal fusion
* discogenic nerve compression or instability (flexion-extension X-ray film shows > 5mm of sagittal-plane translation)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Chinese/English Version Oswestry Disability Index (ODI) | 6 months
  The ODI comprises 10 questions covering areas related to: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, sexual life and traveling.

SECONDARY OUTCOMES:
Pain medication | 6 months
  Dosage of pain medication taken by the participant each day will be recorded.
Duration of hospital stay | 6 months
  The length of hospital stay will be documented
11-point numeric pain rating scale (NPRS) for measuring back/leg pain | 6 months
  The current back/leg pain intensity of each participant will be quantified by an 11-point NPRS, where 0 means no pain and 10 means the worst imaginable pain.
Physical activity monitoring | 6 months
  An ActiGraph sensor will be used to quantify physical activity level of patients before and after surgery at different time points.
The Chinese version of EuroQol-5D-3L for measuring quality of life | 6 months
  The Chinese version of EuroQol-5D-3L questionnaire comprises the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The descriptive system involves 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain has three levels of responses: no problems, some problems, extreme problems. The participant chooses the most appropriate statement in each domain. The EQ VAS quantifies the respondent's perceived health-related quality of life on a vertical VAS where 0 means 'worst imaginable health state', and 100 means 'best imaginable health state'.
Swiss Spinal Stenosis Questionnaire | 6 months
  This self-administered questionnaire comprises 18 questions in three subscales: 6 questions in the symptom severity scale (ranging from 1 to 5), 6 questions in the physical function scale (ranging from 1 to 4), and 6 questions in the patient's satisfaction with treatment scale (ranging from 1 to 4). The result is expressed as a percentage of the maximum possible score. A higher score indicates more disability.
International Physical Activity Questionnaire | 6 months
  International Physical Activity Questionnaire (Chinese short-form version) is a 9-item questionnaire aiming to monitor an individual's leisure-time physical activity, work/transport-related physical activity, and domestic/gardening physical activity over the last 7-day period. Based on the duration, frequency and intensity of the reported physical activity, a person will be classified as physically inactive, minimally active, and health-enhancing physically active.
Clinical Global Impression of Change | 6 months
  The patient's perceived changes immediately after the prehabilitation will be measured by the Clinical Global Impression of Change scale, which is a 7-point numerical rating scale. The value of 1 indicates very much improved, while 7 means very much worse. It will help evaluate the effect of prehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No